CLINICAL TRIAL: NCT04892212
Title: A Pilot Study of Sirolimus in Treatment of Proteinuric Flares of Lupus Nephritis
Brief Title: Sirolimus in Treatment of Proteinuric Flares of Lupus Nephritis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: North China Pharmaceutical Group Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2743
Record Dates: First submitted 2021-05-10; First posted 2021-05-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Lupus Nephritis; Immunosuppression; Effect of Drug
Keywords: Sirolimus; Lupus Nephritis; Renal Flare
MeSH Terms: conditions — Lupus Nephritis | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sirolimus group (Experimental): 1. The initial dose of sirolimus is 1mg/day. And the serum trough level of sirolimus is monitored at Week 2, Week 4, Week 8, and Week 12，respectively. The target serum trough level of sirolimus is 5-8 ng/mL. The dose of sirolimus is titrated according to therapeutic drug level monitoring.
  2. The previous immunosuppressive medication is not allowed to be changed during the 3-month follow-up, unless premature discontinuation from study.
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — The daily dose of sirolimus is divided twice.
  Other Names: Rapamycin

SUMMARY:
This a single-centre, one-arm, open-label pilot study. Eligible patients with mild proteinuric flares of lupus nephritis Class III/IV±V are received sirolimus without changing previous immunosuppressive medication during 12-week follow-up.

Primary Objective:

* To investigate the efficacy of sirolimus for mild proteinuric flares in patients with Class III/IV±V lupus nephritis

Secondary Objective:

* To assess the safety and tolerability of sirolimus treatment for mild proteinuric flares in patients with Class III/IV±V lupus nephritis

DETAILED DESCRIPTION:
Lupus nephritis is a common and serious complication of systemic lupus erythematosus (SLE). It often requires aggressive immunosuppressive therapy. Although majority of patients with severe lupus nephritis achieve a complete or partial remission after 6-month induction treatment, renal flares can still occur during maintenance therapy. Whether patients with mild proteinuric flares should receive intensive immunosuppressive therapy is unclear. In pathogenesis of SLE, T-cell dysfunction is attributed to the activation of the mammalian target of rapamycin (mTOR). Previous prospective and retrospective studies in SLE or lupus nephritis showed the effect of mTOR blockade on systemic disease activity index or severe lupus nephritis as initial or maintenance therapy.

Eligible subjects with biopsy-proven Class III/IV±V lupus nephritis(ISN/RPS 2003) are received oral sirolimus without change previous immunosuppressive therapy. We follow up the included patients at Week 2, Week 4, Week6, Week 8 and Week 12 regularly.

The investigator will actively detect and inquire about the occurrence of adverse events (AEs)/ severe adverse events (SAEs) at every visit/ contact during the study. The clinical trials insurance is prepaid by sponsor to cover the design risks of the protocol and liability/ compensation to the research subject for bodily injury or death resulting from their participation in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven Class III or IV±V lupus nephritis (ISN/RPS 2003 lupus nephritis classification) with biopsy performed within 48 weeks before inclusion.
* Males or females aged 18 to 60 years old at the time of screening.
* The mild proteinuric flare of lupus nephritis is defined as meeting all of the following criteria :

  1. Persistently increased proteinuria after complete remission, and 24-hr proteinuria≥1.0g/day or doubling of proteinuria after partial remission, and 24-hr proteinuria≥2.0g/day
  2. No hypoalbuminemia: serum albumin ≥35g/L
  3. Stable renal function: serum creatinine<25% increase above the level at the time of renal disease remission
* Eligible to sign informed-consent independently

Exclusion Criteria:

* Renal disease unrelated to SLE (e.g. diabetes mellitus, other glomerular or tubulointerstitial diseases, renovascular disease), or transplanted kidney
* Estimate glomerular filtration rate (eGFR by CKD-EPI)<45mL/min per 1.73m^2 at the time of screening
* Renal biopsy showing cellular of fibrocellular crescent in more than 25% of glomeruli
* Central nervous system (CNS) or other severe organ manifestations of lupus that necessitate aggressive immunosuppressive therapy on its own.
* Co-morbidities that require corticosteroid therapy (e.g. asthma, inflammatory bowel disease)
* Any increased dose of corticosteroids or other immunosuppressive medication including cyclophosphamide, mycophenolate, leflunomide, calcineurin inhibitors, azathioprine, methotrexate, or use of biological agents regardless of duration, with the past six months
* Hepatitis B virus (HBV) or Hepatitis C virus (HCV) infection history: seropositivity of HBV surface antigen (HBsAg) or HCV antibodies (HCV-Ab)
* Women who are pregnant or breastfeeding
* Women with childbearing potential or their male partners, who refuse to use an effective birth control method

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-06-30 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
The number of patients achieving sustained Renal Response(RR) | at the end of 12 weeks (3 months) from baseline
  Sustained RR is defined as satisfying all of the following criteria:
  1)Proteinuria is improved by ≥50% compared with baseline
  2)24-hr urine protein < 1g
  3)Serum creatinine is not higher than 15% above baseline level
  4)No occurrence of non-renal disease flare after achieving response to treatment.

SECONDARY OUTCOMES:
Complete renal remission | at the end of 12 weeks (3 months) from baseline
  1. 24-hr urine protein<0.3g/day or urine Protein-Creatinine ratio (uPCR)<300mg/g
  2. Serum creatinine not higher than 15% above baseline level
Partial renal remission | at the end of 12 weeks (3 months) from baseline
  1. 24-hr urine protein<3.5g/day or uPCR<3500mg/g
  2. Serum creatinine not higher than 15% above baseline level
Rate of non-renal flare | during the 3-month follow up
  Central nervous system or other severe organ manifestations of SLE that necessitate aggressive immunosuppressive therapy on its own
Safety and tolerability of study medications | during the 3-month follow up
  The following parameters will be monitored:
  1. Increase of serum creatinine level>15% from baseline and whether it is reversible or irreversible
  2. Episodes with sirolimus level above the target range
  3. New-onset hypertension or worsening hypertensive control that required increase of antihypertensive medication
  4. Infectious requiring hospitalization and the causative agents
  5. Hospitalization episodes- cause, duration (days)
  6. Hypokalemia: serum potassium <3.5mmol/L
  7. Metabolic acidosis with HCO3 <17mmol/L
  8. New-onset hypercholesterolemia present at 3 months or beyond from baseline and/or addition of lipid-lowering drug(s).
  9. Premature discontinuation from the study due to treating intolerance
  10. Premature discontinuation from the study due to rapid disease progression or other reasons
  11. Failure to adhere to the protocol defined corticosteroid reduction regimen
  12. Other adverse clinical events or events considered clinically significant
Increase of serum creatinine level>15% from baseline | during the 3-month follow up
  Increase of serum creatinine level (μmol/L)>15% from baseline and whether it is reversible or irreversible.
Episodes with sirolimus level above the target range | during the 3-month follow up
  Episodes with sirolimus level above the target range（serum sirolimus trough level>8ng/mL) will be recorded.
New-onset hypertension or worsening hypertensive control that required increase of antihypertensive medication | during the 3-month follow up
  Hypertension be diagnosed when a person's systolic blood pressure (SBP) in the office or clinic is ≥140 mm Hg and/or their diastolic blood pressure (DBP) is ≥90 mm Hg following repeated examination.
  New-onset hypertension or worsening hypertensive control that required increase of antihypertensive medication will be recorded.
Infection requiring hospitalization | during the 3-month follow up
  Infection requiring hospitalization will be recorded including the site of infection, the causative agent and duration (days).
Hypokalemia | during the 3-month follow up
  Serum potassium <3.5mmol/L
Hypercholesterolemia | during the 3-month follow up
  New-onset hypercholesterolemia present during follow-up or beyond from baseline and/or addition of lipid-lowering drug(s)
Premature discontinuation from the study | during the 3-month follow up
  The time of of discontinuation from study will be recorded, and the discontinuation is due to:
  1. treating intolerance
  2. rapid disease progression
  3. other reasons
Failure to adhere to the protocol | during the 3-month follow up
  Failure to adhere to the protocol including:
  1. do not titer the dose of sirolimus following study protocol
  2. increase the dose of other immunosuppressives personally without the permission of physician
Changes in Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) | from baseline to end of 12 weeks
  Safety of Estrogens in Lupus Erythematosus National Assessment-Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) assesses disease activity by scoring 24 weighted disease activity descriptors of SLE as "present" or "absent" in preceding 10 days. A patient's total score is the sum of all marked SLE-related descriptors; a total score ranges between 0 and 105, with a higher score representing a more significant degree of disease activity.
  Assessment scales of SELENA-SLEDAI is available online.
Changes in Physician Global Assessement (PGA) | from baseline to end of 12 weeks
  The Physician Global Assessment (PGA) is a visual analog scale (VAS) using 3 benchmarks for assessing disease activity over the last 2 weeks. Mild flare will score 1.0 point, moderate flares will score a 2.0-2.5 point and severe flares will score a 3 on the 0-3 analog scale. PGA is available online.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-mei Li, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yap DYH, Tang C, Chan GCW, Kwan LPY, Ma MKM, Mok MMY, Chan TM. Longterm Data on Sirolimus Treatment in Patients with Lupus Nephritis. J Rheumatol. 2018 Dec;45(12):1663-1670. doi: 10.3899/jrheum.180507. Epub 2018 Oct 1. PMID 30275264
- [Background] Lai ZW, Kelly R, Winans T, Marchena I, Shadakshari A, Yu J, Dawood M, Garcia R, Tily H, Francis L, Faraone SV, Phillips PE, Perl A. Sirolimus in patients with clinically active systemic lupus erythematosus resistant to, or intolerant of, conventional medications: a single-arm, open-label, phase 1/2 trial. Lancet. 2018 Mar 24;391(10126):1186-1196. doi: 10.1016/S0140-6736(18)30485-9. Epub 2018 Mar 15. PMID 29551338
- [Background] Eriksson P, Wallin P, Sjowall C. Clinical Experience of Sirolimus Regarding Efficacy and Safety in Systemic Lupus Erythematosus. Front Pharmacol. 2019 Feb 6;10:82. doi: 10.3389/fphar.2019.00082. eCollection 2019. PMID 30787878
- [Background] Esatoglu SN, Seyahi E. Is sirolimus a treatment option for patients with systemic lupus erythematosus? Clin Exp Rheumatol. 2019 Nov-Dec;37 Suppl 122(6):13. Epub 2019 Jul 12. No abstract available. PMID 31376256
- [Background] Ma MKM, Yung S, Chan TM. mTOR Inhibition and Kidney Diseases. Transplantation. 2018 Feb;102(2S Suppl 1):S32-S40. doi: 10.1097/TP.0000000000001729. PMID 29369972